CLINICAL TRIAL: NCT00293774
Title: A Provincial Initiative to Examine the Efficacy, Cost-effectiveness and Long-term Safety of Alternative Hip Bearing Surfaces Versus Conventional Therapy for Degenerative Joint Disease of the Hip
Brief Title: Alberta Hip Improvement Project
Status: Completed | Type: Observational
Sponsor: Alberta Bone and Joint Health Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ABHIP-00001
Record Dates: First submitted 2006-02-16; First posted 2006-02-20 (Estimated); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Arthroplasty, Replacement, Hip
Keywords: Prospective; Conventional therapy; Registry; Metal-on-metal; Ceramic-on-ceramic; Hip Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples retained for cobalt and chromium metal ion level analysis on select cohort.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Standard: Standard hip replacement subjects (polyethylene)
- Alternative Bearing: Subjects with ceramic on ceramic total hip replacement or metal on metal hip resurfacing.

SUMMARY:
A study to determine the effectiveness and safety of the use of metal-on-metal hip resurfacing (for example the birmingham hip) when compared to conventional total hip replacement.

DETAILED DESCRIPTION:
This study is designed to provide orthopedic surgeons and decision makers with evidence-based health measures for patients that are treated by orthopedic surgeons for degenerative joint disease of the hip in Alberta. This study is provincial initiative to determine whether new alternative hip bearing surfaces improve patient outcomes and/or decrease health resource utilization in patients with degenerative joint disease of the hip in Alberta. The primary objective is to compare time to revision for patients receiving alternative hip bearing surfaces to patients receiving conventional total hip replacements. Secondary objectives are to evaluate long-term safety; to evaluate costs; to determine if alternative hip bearing surfaces improve patient function; to develop evidence base guidelines for the implementation of alternative hip bearing surfaces in Alberta; do develop a modal to assess other technologies and health advances; to develop an Alberta HIP registry

ELIGIBILITY:
Inclusion Criteria:

* documentation of DJD of hip
* patient at least 18 years
* patient able to provide written consent
* Male under 65 years, female under 56 years
* Orthopedic surgeon has received appropriate training to implant an alternative device

Exclusion Criteria:

* renal failure (MOM only)
* child bearing potential (MOM only)
* inappropriate femoral anatomy, including evidence of osteoporosis
* inflammatory arthritis (MOM)
* Unwilling to consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males between the ages of 18-65 and females between the ages of 18-55
Sampling Method: Probability Sample
Enrollment: 1632 (Actual)
Dates: Start 2004-06; Primary Completion 2011-01 (Actual); Study Completion 2021-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James MacKenzie, M.D., Principal Investigator — University of Calgary; Greg O'Connor, MD, Principal Investigator — University of Alberta
Locations (1):
- Alberta Bone and Joint Health Institute, Calgary, Alberta, Canada